CLINICAL TRIAL: NCT04702048
Title: The Evaluation of Retinal PhotoReceptors And Vasculature in Moderate and Severe Non-proliferative Diabetic Retinopathy Patients After Intravitreal Aflibercept on Using Adaptive Optics Imaging Study (PRAVA) Study
Brief Title: Evaluation of the Retina in Patients With Non-proliferative Diabetic Retinopathy After Aflibercept Injection in the Eye
Acronym: PRAVA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: sponsor withdrew funding
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jesse Schallek, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005589
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Retinopathy, Diabetic
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aflibercept injection (Experimental): Intravitreal injection of Aflibercept
  Interventions: Drug: Aflibercept Injection
- Sham injection (Placebo Comparator): Empty syringe with no needle
  Interventions: Drug: Sham injection

INTERVENTIONS:
Drug: Aflibercept Injection — Patients randomized to Arm A will receive 2 mg IVT aflibercept injections every 4 weeks (Q4W) to Week 20, followed by 2-mg aflibercept injections Q8W to Week 52.
  Arms: Aflibercept injection
Drug: Sham injection — Patients randomized to Arm B will receive sham intravitreal injections every 4 weeks (Q4W) to Week 20, followed by sham intravitreal injections Q8W to Week 52. Sham means eye will be numbed and a syringe with no needle will be touched to the eye.
  Arms: Sham injection

SUMMARY:
The purpose of this study is to specifically assess the effect of intravitreal aflibercept injections on the health of cells and the flow of blood through the retinal blood vessels by using advanced technology called adaptive optics.

ELIGIBILITY:
Inclusion Criteria:

* Documented Type 1 or 2 diabetes mellitus who have moderately severe to severe NPDR (DRSS levels 47 or 53) as confirmed by 2 independent physician evaluators.
* Age ≥18 years
* Willingness and the ability to provide signed informed consent, comply with clinic visits and study-related procedure, and provide Health Insurance Portability and Accountability Act authorization
* BCVA of ≥ 73 letters, inclusive (≥20/40 approximate Snellen equivalent), using the ETDRS protocol at the initial testing distance of 4 meters (see the BCVA manual for additional details) on Day 1
* Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good quality CFPs (including ETDRS 7 modified fields or Optos ultra-widefield image to permit grading of diabetic retinopathy and assessment of the retina) and other imaging modalities, including AOSLO.
* No center-involved macular edema (defined as fluid within 1000 microns of the fovea)
* HbA1c of ≤10% within 2 months prior to the first injection visit date
* For men* and women** of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the final dose of study treatment. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly. Contraception is not required for men with documented vasectomy. Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Exclusion Criteria:

* Presence of DME threatening the center of the macula (within 1,000 microns of the foveal center) in the study eye
* Evidence of retinal neovascularization on clinical examination or FA
* Any prior focal or grid laser photocoagulation (within 1,000 microns of the foveal center) or any prior PRP in the study eye
* Any prior systemic anti-VEGF treatment or IVT anti-VEGF treatment in the study eye
* Any prior intraocular steroid injection in the study eye
* History of vitreoretinal surgery in the study eye
* Intraocular pressure (IOP) ≥25 mm Hg in the study eye
* Evidence of active infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye
* Any intraocular inflammation or infection in either eye within 3 months of the screening visit
* Current Anterior segment neovascularization, vitreous hemorrhage, or tractional retinal detachment visible at the screening assessments in the study eye
* Ocular media of insufficient quality to obtain fundus and optical coherence tomography (OCT), and adaptive optics images in the study eye
* Hemoglobin A1c (HbA1c) >12%, or if HbA1c is ≤12%, diabetes mellitus is uncontrolled in the opinion of the investigator
* Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of IVT injections, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety
* Uncontrolled blood pressure (defined as systolic >160 mm Hg or diastolic >95 mm Hg while patient is sitting)
* History of cerebrovascular accident or myocardial infarction within 6 months of day 1
* Renal failure, dialysis, or history of renal transplant
* Positive serum hCG/urine pregnancy test at the screening or baseline visit
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk for treatment complications
* Participation as a patient in any interventional ocular clinical study within the 12 weeks prior to day 1 of the study
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception prior to the initial dose/start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly. Contraception is not required for men with documented vasectomy.

Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in photoreceptor mosaic | baseline to 52 weeks
  Adaptive optics imaging will be used to visualize the photoreceptor cells in the eye and the number of photoreceptor cells will be quantified at baseline and 52 weeks.
Mean change in photoreceptor cell density | baseline to 52 weeks
  Adaptive optics imaging will be used to visualize the photoreceptor cells in the eye and the number of photoreceptor cells per square micron of image will be quantified at baseline and 52 weeks.
Mean change in photoreceptor cell spacing | baseline to 52 weeks
  Adaptive optics imaging will be used to visualize the photoreceptor cells in the eye and a measurement of the space between photoreceptor cells will be calculated at baseline and 52 weeks.

SECONDARY OUTCOMES:
Percent of participants with any ocular adverse events | 52 weeks
Percent of participants with a severe ocular adverse events | 52 weeks
Percent of participants with a non-ocular adverse events | 52 weeks
Percent of participants with a severe non-ocular adverse events | 52 weeks
Mean change in foveal avascular zone area | baseline to 52 weeks
  Adaptive optics and optical coherence tomography angiography will be used to quantify the area of the macula without blood vessels.
Mean change in macular retina non-perfusion area | baseline to 52 weeks
  Optical coherence tomography angiography will be used to quantify the area of the macula without blood vessels.
Mean change in capillary blood cell velocity | baseline to 52 weeks
  Adaptive optics will be used to quantify the mean speed of blood cells passing through the retinal blood vessels.
Mean change in blood cell flux | baseline to 52 weeks
  Adaptive optics will be used to quantify the mean number o blood cells passing through the blood vessel per period of time.
Mean change in number of capillary occlusions | baseline to 52 weeks
  Adaptive optics will be used to quantify the number of time blood flow stops (occlusions) in the eye blood vessels.
Change in duration of capillary occlusions | baseline to 52 weeks
  Adaptive optics will be used to quantify the length of time blood flow stops (occlusions) in the eye blood vessels.
Proportion of patients with a ≥ 2-step DRS improvement from baseline on the Early Treatment Diabetic Retinopathy Study Diabetic Retinopathy Severity Scale (ETDRS DRSS) | 52 weeks
  The ETDRS DRSS measures the number of vascular changes seen in the eye due to diabetes. The range is 10-81. A lower value indicates a better health outcome. The steps cut offs are 10, 20, 35, 43, 47, 53, 60, 61, 65, 71, 75, 81.
Proportion of patients with a ≥ 3-step DRS improvement from baseline on the ETDRS DRSS. | 52 weeks
  The ETDRS DRSS measures the number of vascular changes seen in the eye due to diabetes. The range is 10-81. A lower value indicates a better health outcome. The steps cut offs are 10, 20, 35, 43, 47, 53, 60, 61, 65, 71, 75, 81.
Proportion of participants developing a vision-threatening complication due to diabetic retinopathy | 52 weeks
  Progression to proliferative diabetic retinopathy, develop of diabetic macular edema, development of neovascular glaucoma and vitrous hemorrhage are all vision-threatening complications.
Mean change in central subfield thickness | baseline to 52 weeks
  Optical coherence tomography will be used to measure the central subfield thickness.
Proportion of patients with absence of intraretinal fluid | 52 weeks
  Optical coherence tomography will be used to measure presence or absence of intraretinal fluid.
Proportion of patients with absence of subretinal fluid | 52 weeks
  Optical coherence tomography will be used to measure presence or absence of intraretinal fluid.
Mean change in mean parafoveal macular ganglion cell layer and inner plexiform layer (mGCIPL) thickness | baseline to 52 weeks
  Optical coherence tomography will be used to measure mGCIPL thickness.
Mean change in Best Corrected Visual Acuity (BCVA) | baseline to 52 weeks
  BCVA is a visual test using letters and change will be measured as the number of letters correctly read.
Change in proportion of patients with BCVA Snellen equivalent of 20/40 or better | baseline to 52 weeks
Proportion of participants who receive panretinal photocoagulation (PRP) | week 52
  PRP is a laser procedure for proliferative diabetic retinopathy that will be performed based on clinical evaluation of the patient.
Proportion of participants who receive intravitreal aflibercept | week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Flaum Eye Institute, University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided